CLINICAL TRIAL: NCT00559273
Title: An Open-label, Randomized, Multicenter, Parallel-group Study to Demonstrate Correction of Anemia Using Once Every 4 Weeks Subcutaneous Injections of RO0503821 in Patients With Chronic Kidney Disease Who Are Not on Dialysis
Brief Title: A Study of Subcutaneous Mircera Once Monthly in the Treatment of Anemia in Participants With Chronic Kidney Disease Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH20052
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Renal Anemia, Chronic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — continuous erythropoietin receptor activator; Darbepoetin alfa

ARMS (2):
- Mircera (Experimental): Participants will receive Mircera (Methoxy polyethylene glycol-epoetin beta), administered subcutaneously (SC) at a starting dose of 1.2 mcg/kg once every 4 weeks for 28 weeks.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta
- Darbepoetin Alfa (Active Comparator): Participants will receive darbepoetin alfa, administered SC once weekly or once every 2 weeks according to local labeling specifications for 28 weeks.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — 1.2 mcg/kg SC monthly, starting dose
  Other Names: Mircera; RO0503821
  Arms: Mircera
Drug: Darbepoetin alfa — 0.45 mcg/kg SC weekly or 0.75 mcg/kg every 2 weeks, starting dose
  Arms: Darbepoetin Alfa

SUMMARY:
This study will compare the efficacy and safety of subcutaneous Mircera and subcutaneous darbepoetin in the treatment of renal anemia in participants with chronic kidney disease who are not on dialysis and not receiving erythropoiesis-stimulating agents (ESA). Participants will be randomized to receive either Mircera once every 4 weeks, at a starting dose of 1.2 micrograms/kilogram (mcg/kg), or darbepoetin alfa once weekly, at a starting dose of 0.45 mcg/kg (or once every two weeks, 0.75 mcg/kg). The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic kidney disease (CKD) stage 3 (creatinine clearance [CrCl]/ glomerular filtration rate [GFR] 30 to 59 milliliter per minutes per 1.73 meter square [mL/min/1.73m^2]) or Stage 4 (CrCl/GFR 15-29 mL/min/1.73m^2) who did not require dialysis. CrCl/GFR was estimated with the Cockcroft-Gault equation or the abbreviated Modification of Diet in Renal Disease (MDRD) equation
* Anemia defined as baseline Hb concentration less than (<) 10.5 gram per deciliter (g/dL)

Exclusion Criteria:

* Previous therapy with any ESA within 12 weeks prior to screening
* Renal allograft in place
* Immunosuppressive therapy in the 12 weeks prior to screening
* Overt gastrointestinal bleeding and red blood cells (RBC) transfusions within 8 weeks before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (64):
- Australia (5):
  - Adelaide
  - Clayton
  - Gosford
  - Parkville
  - Reservoir
- Belgium (2):
  - Aalst
  - Roeselare
- Canada (4):
  - Edmonton, Alberta
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (6):
  - Cahors
  - Clermont-Ferrand
  - Limoges
  - Lyon
  - Nice
  - Paris
- Germany (4):
  - Berlin
  - Bonn
  - Heilbronn
  - Homburg/saar
- Greece (4):
  - Alexandroupoli
  - Larissa
  - Thessaloniki
  - Volos
- Hong Kong, Hong Kong
- Hungary (5):
  - Baja
  - Budapest
  - Esztergom
  - Hatvan
  - Szigetvár
- Israel (3):
  - Haifa
  - Kfar Saba
  - Petah Tikva
- Italy (6):
  - Como
  - Lecco
  - Lodi
  - Mestre
  - Modena
  - Pavia
- Poland (10):
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Radom
  - Rzeszów
  - Sieradz
  - Szczecin
  - Warsaw
  - Wroclaw
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Saratov
- Seoul, South Korea
- Spain (5):
  - Barcelona
  - Madrid
  - Palma de Mallorca
  - Seville
  - Valencia
- Taiwan (2):
  - Taichung
  - Taipei
- Thailand (3):
  - Bangkok
  - Nakhon Ratchasima
  - Pathum Thani

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera: Participants received Mircera (Methoxy polyethylene glycol-epoetin beta), administered subcutaneously (SC) at a starting dose of 1.2 microgram per kilogram (mcg/kg) once every 4 weeks for 28 weeks.
- Darbepoetin Alfa: Participants received darbepoetin alfa, administered SC once weekly or once every 2 weeks according to local labeling specifications for 28 weeks.
Period: Correction Period (20 Weeks)
Arm/Group | Mircera | Darbepoetin Alfa
Started | 153 | 154
Treated | 151 | 154
Completed | 144 | 142
Not Completed | 9 | 12
Not completed — Death | 3 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Participant treated by another center | 0 | 1
Not completed — Did not received study treatment | 2 | 0
Period: Evaluation Period (8 Weeks)
Arm/Group | Mircera | Darbepoetin Alfa
Started | 144 | 142
Completed | 141 | 137
Not Completed | 3 | 5
Not completed — Death | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study medication and attended safety follow-up, whether they withdrew prematurely or not. Participants were assigned to the treatment group as treated. One participant randomized to Mircera, received darbepoetin alfa and included in darbepoetin alfa arm.
Groups:
- Mircera: Participants received Mircera (Methoxy polyethylene glycol-epoetin beta), administered SC at a starting dose of 1.2 mcg/kg once every 4 weeks for 28 weeks.
- Total: Total of all reporting groups
Arm/Group | Mircera | Darbepoetin Alfa | Total
Number analyzed (Participants) | 150 | 155 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (14.37) | 67.4 (13.40) | 66.3 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 87 | 172
  Male | 65 | 68 | 133

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemoglobin (Hb) Response
Description: Hb response was an observed increase in Hb greater than or equal to (>=) 1.0 gram per deciliter (g/dL) from baseline and an Hb concentration >= 10.0 g/dL before the end of the study without red blood cells (RBC) transfusion before response.
Time Frame: Baseline up to Week 28
Population: Intent-to-treat (ITT) population included all randomized participants. Participants were analyzed according to the study treatment assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 153 | 154
percentage of participants | 94.12 [89.13 to 97.28] | 93.51 [88.38 to 96.84]
Statistical Analysis 1: Comparison: Mircera; The p-value was the probability that the number of responders is greater than or equal to the observed number, although the true response rate was smaller or equal to 60%. Null hypothesis (H0): p-value <=0.6; alternate hypothesis (H1): p-value >0.6; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Darbepoetin Alfa; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Change in Hemoglobin (Hb) Concentration Between Baseline and Evaluation Period
Description: A time adjusted average baseline Hb concentration was calculated using the trapezoid rule from all available Hb measurements taken during the baseline period. The average evaluation period Hb concentration for each individual was calculated using the same method, from all their available measurements taken during the 2 month evaluation period (Week 21 to 28). The change in Hb concentration between the baseline and evaluation period was calculated by subtracting the baseline Hb from the evaluation period Hb. All blood samples for Hb measurements were taken prior to study drug administration.
Time Frame: Baseline (measurements at Week -2, Week -1 and Day 1) and Evaluation Period (Week 22, Week 24, Week 26, Week 28)
Population: ITT population. Here, N (number of participants analyzed)=participants evaluable for this measure. Missing data were imputed using last value carried forward.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 150 | 151
g/dL | 1.66 (1.18) | 1.69 (0.95)
Statistical Analysis 1: Comparison: Mircera vs Darbepoetin Alfa; Test type: Non-Inferiority or Equivalence — MIRCERA treatment was regarded as non-inferior to the darbepoetin alfa reference group if the lower limit of the CI was greater than -0.75 g/dL; p < 0.0001, ANCOVA; Adjusted Mean Difference = -0.036, 95% CI 2-sided [-0.252 to 0.180], Standard Error of Mean 0.1097

3. Secondary Outcome: Hemoglobin (Hb) Concentration Over the Time
Description: The hemoglobin concentration was measured in g/dL every 2 weeks and at final visit.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and final visit (Week 29)
Population: ITT population. Here, n=number of evaluable participants at specified time point, respectively for each group.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 153 | 154
g/dL
  Baseline (n=153, 154) | 9.53 (0.74) | 9.53 (0.65)
  Week 2 (n=149, 151) | 10.22 (0.91) | 10.14 (0.93)
  Week 4 (n=149, 148) | 10.37 (1.17) | 10.74 (1.02)
  Week 6 (n=149, 148) | 10.94 (1.23) | 11.28 (1.08)
  Week 8 (n=148, 147) | 11.08 (1.29) | 11.74 (1.05)
  Week 10 (n=150, 146) | 11.36 (1.27) | 11.78 (1.02)
  Week 12 (n=149, 145) | 11.24 (1.17) | 11.82 (1.03)
  Week 14 (n=145, 143) | 11.53 (1.11) | 11.81 (1.04)
  Week 16 (n=144, 145) | 11.50 (1.16) | 11.76 (1.06)
  Week 18 (n=144, 141) | 11.41 (1.04) | 11.45 (0.94)
  Week 20 (n=142, 140) | 11.14 (0.92) | 11.34 (0.81)
  Week 22 (n=142, 138) | 11.39 (1.02) | 11.43 (0.86)
  Week 24 (n=140, 140) | 11.06 (0.98) | 11.26 (1.00)
  Week 26 (n=139, 136) | 11.17 (0.96) | 11.24 (0.94)
  Week 28 (n=139, 136) | 11.08 (0.97) | 11.48 (0.91)
  Week 29 (n=151, 151) | 11.07 (1.10) | 11.31 (1.12)

4. Secondary Outcome: Time to Hemoglobin Response
Description: Time to Hb response is defined as the number of study days until the first occurrence of an Hb response. Participants without events were censored at the time of evaluation. Median and 95 percent (%) confidence interval (CI) were estimated using Kaplan-Meier Survival Analysis. Hb response was an observed increase in Hb >=1.0 g/dL from baseline and an Hb concentration >= 10.0 g/dL before the end of the study without RBC transfusion before response.
Time Frame: Baseline up to Week 28
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 153 | 154
days | 43 [37 to 43] | 29 [29 to 41]

5. Secondary Outcome: Percentage of Participants With Red Blood Cell (RBC) Transfusions
Description: The percentage of participants who received RBC transfusions during the titration and evaluation periods were reported.
Time Frame: Baseline up to Week 28
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 153 | 154
percentage of participants | 3.3 | 6.5

6. Secondary Outcome: Percentage of Participants Who Had at Least 1 Hemoglobin Value Exceeding 12.0 g/dL
Description: Percentage of participants having at least one Hb value greater than (>) 12 g/dL during the first 8 weeks of the study was reported.
Time Frame: Baseline to Week 8
Population: ITT population. Here, N=number of participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 151 | 151
percentage of participants | 25.8 | 47.7

7. Secondary Outcome: Percentage of Participants With Stable Hemoglobin Response
Description: A participant was defined as having achieved a stable Hb response, if at least 75 percent (%) of the scheduled Hb values were between 10.0 g/dL and 12.0 g/dL and >=1.0 g/dL from baseline for any 8-week time period, regardless of the requirement for dose adjustment for Hb maintenance. Achievement of stable response was determined using a moving 8-week time window, moving forward by 14 days in each iteration starting at Day 15, searching to see if the following conditions were met: 1) At least 3 scheduled Hb values (75% of the scheduled Hb values) in any 8-week time window were >=1.0 g/dL from baseline (as calculated above) and within the range of 10.0 g/dL to 12.0 g/dL. 2). There were at least 3 recorded Hb values within the time window.
Time Frame: Baseline to Week 28
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 153 | 154
percentage of participants | 68.63 [60.64 to 75.88] | 72.73 [64.97 to 79.58]

8. Secondary Outcome: Percentage of Participants Who Required Dose Adjustments to Achieve a Stabilized Response
Description: The total number of dose adjustments needed to achieve stabilized response was calculated from Day 1 until the first 8-week time window in which response was achieved. A participant was defined as having achieved a stable Hb response, if at least 75% of the scheduled Hb values were between 10.0 g/dL and 12.0 g/dL and >=1.0 g/dL from baseline for any 8-week time period, regardless of the requirement for dose adjustment for Hb maintenance. Achievement of stable response was determined using a moving 8-week time window, moving forward by 14 days in each iteration starting at Day 15, searching to see if the following conditions were met: 1) At least 3 scheduled Hb values (75% of the scheduled Hb values) in any 8-week time window were >=1.0 g/dL from baseline (as calculated above) and within the range of 10.0 g/dL to 12.0 g/dL. 2) There were at least 3 recorded Hb values within the time window.
Time Frame: Baseline to Week 28
Population: ITT population. Here, N=number of participants analyzed for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 105 | 112
percentage of participants
  Dose Increase(s) only | 41.9 | 18.8
  Dose Decrease(s) only | 8.6 | 19.6
  Dose Decrease(s) and Increase(s) | 11.4 | 18.8
  No Dose Change | 38.1 | 42.9

ADVERSE EVENTS:
Time Frame: Baseline up to 29 weeks
Description: Safety population included all randomized participants who received at least 1 dose of study medication and attended safety follow-up, whether they withdrew prematurely or not. Participants were assigned to the treatment group as treated. One participant randomized to Mircera, received darbepoetin alfa and included in darbepoetin alfa arm.
Arm/Group | Mircera | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 28/150 | 39/155
Other Adverse Events (participants affected / at risk) | 50/150 | 65/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=150) | Darbepoetin Alfa (N=155)
Renal impairment (Renal and urinary disorders) | 4 | 9
Azotaemia (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 1
Diabetic gangrene (Infections and infestations) | 1 | 0
Meningoencephalitis bacterial (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Starvation (Metabolism and nutrition disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penis carcinoma metatstatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Sudden death (General disorders) | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=150) | Darbepoetin Alfa (N=155)
Hypertension (Vascular disorders) | 24 | 37
Hypotension (Vascular disorders) | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 9 | 11
Nasopharyngitis (Infections and infestations) | 5 | 8
Constipation (Gastrointestinal disorders) | 5 | 12
Diarrhoea (Gastrointestinal disorders) | 10 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.